CLINICAL TRIAL: NCT06596668
Title: An Open-Label, Phase 1 Study to Characterize the Effects of a Strong Cytochrome P450 3A4 Inducer on the Pharmacokinetics of Bomedemstat in Healthy Adult Participants
Brief Title: Drug-Drug Interaction Study of Bomedemstat and Carbamazepine in Healthy Adult Participants (MK-3543-020)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3543-020; MK-3543-020 (Other: MSD)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — bomedemstat; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bomedemstat + Carbamazepine (Experimental): A single dose of bomedemstat will be administered On Day 1 of Period 1. There will be a washout of 7 days between bomedemstat dosing in Period 1 and the first carbamazepine (CBZ) dose in Period 2. In Period 2, CBZ will be administered twice daily (BID) for 17 consecutive days, with a single dose of bomedemstat coadministered with the morning dose on Day 14.
  Interventions: Drug: bomedemstat; Drug: carbamazepine

INTERVENTIONS:
Drug: bomedemstat — Oral tablet
  Other Names: MK-3543
Drug: carbamazepine — Oral extended-release capsule

SUMMARY:
Researchers have designed a study medicine called bomedemstat (MK-3543) as a new way to treat certain rare blood diseases.

The purpose of this study is to learn what happens to bomedemstat in a person's body over time (a pharmacokinetic or PK study). Researchers will compare what happens to bomedemstat in the body when it is given alone and after multiple doses of another medicine called carbamazepine (CBZ).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months before entering the study.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m^2
* Medically healthy with no clinically significant medical history

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History or presence of any of the following:

  * Seizures
  * Negative reactions in the blood system to any drugs
  * Depression, unusual changes in mood or behavior or suicidal thoughts or behavior
* History of cancer
* Regular user of cannabis products within 6 months before entering the study.
* Unable to stop using or anticipates the use of any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days before entering the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from 0 to infinity (AUC0-inf) of bomedemstat | Predose and at designated timepoints up to 168 hours postdose
  AUC0-inf for bomedemstat in plasma will be determined

SECONDARY OUTCOMES:
Number of participants who experience one or more adverse events (AEs) | Up to approximately 66 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study treatment due to an AE | Up to approximately 25 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Area under the concentration versus time curve from 0 to the time of the last quantifiable sample (AUC0-last) of bomedemstat | Predose and at designated timepoints up to 168 hours postdose
  AUC0-last for bomedemstat in plasma will be determined
Area under the concentration versus time curve from 0 to 24 hours after dosing (AUC0-24) of bomedemstat | Predose and at designated timepoints up to 24 hours postdose
  AUC0-24 for bomedemstat in plasma will be determined
Maximum observed concentration (Cmax) of bomedemstat | Predose and at designated timepoints up to 168 hours postdose
  Cmax for bomedemstat in plasma will be determined
Maximum observed concentration 24 hours after dosing (C24) bomedemstat | Predose and at designated timepoints up to 24 hours postdose
  Cmax for bomedemstat in plasma will be determined
Time to maximum concentration (Tmax) of bomedemstat | Predose and at designated timepoints up to 168 hours postdose
  Tmax for bomedemstat in plasma will be determined
Apparent terminal half-life (t1/2) of bomedemstat | Predose and at designated timepoints up to 168 hours postdose
  t1/2 for bomedemstat in plasma will be determined
Apparent clearance (CL/F) of bomedemstat | Predose and at designated timepoints up to 168 hours postdose
  CL/F for bomedemstat in plasma will be determined
Apparent volume of distribution during terminal phase (Vz/F) of bomedemstat in plasma | Predose and at designated timepoints up to 168 hours postdose
  Vz/F for bomedemstat in plasma will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion, Inc. ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/